CLINICAL TRIAL: NCT06449066
Title: Infectious Complications Associated With the Use of Peri-partum Neuraxial Anaesthesia in Patients With Primary Immunodeficiencies
Brief Title: Primary Immunodeficiencies and Obstetrical Neuraxial Anaesthesia
Acronym: ANEU-DIP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240481
Record Dates: First submitted 2024-05-30; First posted 2024-06-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Infectious Complications (Epidural Abscess or Meningitis); Obstetrical Neuraxial Anaesthesia
Keywords: Primary immunodeficiencies; Neuraxial anaesthesia; Obstetrical anaesthesia; Epidural abscess; Meningitis
MeSH Terms: conditions — Epidural Abscess; Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: CEREDIH (centre de reference des deficits immunitaires héréditaires) cohort Female patients, alive and > 18 years old, registered at the CEREDIH who gave birth in an APHP maternity
  Interventions: Other: Non applicable

INTERVENTIONS:
Other: Non applicable — Non applicable (data collection)

SUMMARY:
The purpose of this study is to evaluate if neuraxial anesthesia (epidural or intradural anesthesia) used during childbirth is associated with more frequent infectious complications in patients with primary immunodeficiencies (PID).

DETAILED DESCRIPTION:
Neuraxial anaesthesia (epidural or intradural) is often used to alleviate pain during labour and childbirth. Although extremely efficient and safe, rare but serious infectious complications such as epidural abscess or meningitis can occur afterwards.

Patients with PID tend to have a greater risk of infectious complications than the general population. With the progress of medical care in those pathologies, female patients are now giving birth more often. The use of neuraxial anaesthesia and the associated infectious complications have never been studied in this population.

The investigators intend to review the medical records of PID patients who gave birth in an APHP hospital in the last 10 years to evaluate the use of neuraxial anesthesia and the frequency of infectious complications associated with neuraxial anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Female patient included in the CEREDIH national register
* Aged > 18 years

Exclusion Criteria:

* Refuse to participate
* Deceased
* Minor
* under judicial protection
* obstetric file not available

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female eligible patients from the CEREDIH cohort will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Number of participants who develop a local or systemic infection, such as an epidural abscess or meningitis, within 28 days after receiving neuraxial anesthesia during delivery | 28 days post-partum
  Occurrence of a local or systemic infection post-neuraxial anesthesia within 28 days after delivery / Infectious complication after obstetrical neuraxial anesthesia / Epidural abscess or meningitis after neuraxial anesthesia

SECONDARY OUTCOMES:
Frequency of Alternative Pain Relief Methods Utilized Due to Contraindications Linked to Primary Immunodeficiency | During labour
  Use of an alternate method for pain-relief during childbirth / Use of another method of pain relief due to a contraindication linked to primary immunodeficiency
Rate of Antibioprophylaxis Administration During Neuraxial Anesthesia | up to 24 hours after birth
  Use of a antibioprophylaxis when performing neuraxial anesthesia
Number of cases where maternity anesthetists identify contraindications to performing neuraxial anesthesia in patients with primary immunodeficiency | During labour
  Possible occurrence of contraindications identified by the maternity anesthetist to the performance of neuraxial anesthesia linked to primary immunodeficiency

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Charlier-Woerther, Principal Investigator — APHP
Locations (1):
- Infectiology mobile team - Department of Infectious and Tropical Diseases, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Beloeuvre A, Anselem O, Tazi A, Keita-Meyer H, Mahlaoui N, Charlier C. Anesthetic management of women with primary immunodeficiencies in the obstetric setting: A French cohort study (ANEU-DIP). J Allergy Clin Immunol Glob. 2025 Jan 30;4(2):100433. doi: 10.1016/j.jacig.2025.100433. eCollection 2025 May. PMID 40226770